CLINICAL TRIAL: NCT04548869
Title: An Open Label, Phase 1 Single Dose Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of CDX-0159 as Add on Therapy in Patients With Cold Contact Urticaria, Symptomatic Dermographism and Cholinergic Urticaria
Brief Title: A Single Dose Study of the Safety, Pharmacokinetics and Pharmacodynamics of CDX-0159 in Patients With Cold Contact Urticaria, Symptomatic Dermographism, or Cholinergic Urticaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX0159-03; 2020-002792-35 (EudraCT Number)
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Cold Urticaria; Cold Contact Urticaria; Symptomatic Dermographism; Symptomatic Dermatographism; Cholinergic Urticaria
MeSH Terms: conditions — Cold Urticaria; Familial dermographism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CDX-0159 (Experimental): 20 patients with Cold Contact Urticaria, 10 patients with Symptomatic Dermographism, and 10 patients with Cholinergic Urticaria will be enrolled and treated with a single dose of CDX-0159
  Interventions: Drug: CDX-0159

INTERVENTIONS:
Drug: CDX-0159 — Administered intravenously

SUMMARY:
This is a study to determine the safety of CDX-0159 in patients with Cold Contact Urticaria, Symptomatic Dermographism, or Cholinergic Urticaria.

DETAILED DESCRIPTION:
This study is an open label Phase 1 study evaluating the safety, pharmacokinetics, and pharmacodynamics of a single dose of CDX-0159 in patients with Cold Contact Urticaria, Symptomatic Dermographism, or Cholinergic Urticaria who remain symptomatic despite treatment with antihistamines. Twenty patients with Cold Contact Urticaria, ten patients with Symptomatic Dermographism, and ten patients with Cholinergic Urticaria will be enrolled in four separate cohorts for a total of 40 patients.

Prospective patients will be screened with tests in clinic as well as daily at home diaries for 2 weeks prior to enrollment. CDX-0159 will be administered intravenously on Day 1. Post-treatment, patients will be followed for 12 weeks with an optional longer term follow up period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of Cold Contact Urticaria, Symptomatic Dermographism, or Cholinergic Urticaria which does not respond to antihistamines

   * Diagnosis for ≥ 3 months; symptoms of both hive (wheal) and itch/burning/painful sensation despite concurrent use of anti-histamines
   * During screening, in clinic, for Cold Contact Urticaria, patients must have a positive cold stimulation test, for Symptomatic Dermographism, patients must have a positive FricTest®, and for Cholinergic Urticaria, patients must have a positive pulse-controlled ergometry (PCE) provocation test
   * On stable dose of antihistamines
2. Other than a diagnosis of Cold Contact Urticaria, Symptomatic Dermographism, or Cholinergic Urticaria, no other conditions which would introduce additional risk factors or would interfere with the study procedures, as determined by the investigator, based on a medical evaluation
3. Female and male patients must use highly effective contraception from the time of the screening visit and for at least 150 days after receipt of study treatment
4. Willing and able to comply with all study requirements and procedures including completion of a daily medication diary and questionnaires

Key Exclusion Criteria:

1. A clearly defined diagnosis of hives or angioedema other than chronic urticaria.
2. Receipt of prior biologic therapy (e.g.: omalizumab, dupilumab, ligelizumab) within past 3 months
3. Treatment with immunosuppressives (e.g. systemic corticosteroids, cyclosporine, methotrexate, dapsone, cyclophosphamide, tacrolimus and mycophenolate mofetil, hydroxychloroquine or others) within 4 weeks or 5 half lives
4. Active COVID-19 infection
5. HIV, hepatitis B or hepatitis C infection

There are additional criteria that your study doctor will review with you to confirm you are eligible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by the incidence and severity of adverse events | From Day 1 through week 12
  Safety of a single dose of CDX-0159 as determined by adverse events

SECONDARY OUTCOMES:
For patients with Cold Contact Urticaria, Change in Critical Temperature Thresholds (CTT) | From Day 1 to Day 85
  The change from baseline in critical temperature thresholds over time as determined by provocation testing using the TempTest®
For patients with Symptomatic Dermographism, change in provocation thresholds | From Day 1 to Day 85
  The change from baseline in provocation thresholds over time as determined by provocation testing using the FricTest®
For patients with Cholinergic Urticaria, changes in baseline Urticaria Activity Score Provocation (UASprovo) | From Day 1 to Day 85
  Changes from baseline and percentage of responders as measured by UASprovo
Changes from baseline in Urticaria Control Test (UCT) | From Day 1 to Day 85
  Changes from baseline and percentage of responders for the UCT and modified UCT
Blood Biomarkers | From Day 1 to Day 85
  Pre-treatment and post-treatment blood samples will be collected and analyzed for changes in Stem Cell Factor
Blood Biomarkers | From Day 1 to Day 85
  Pre-treatment and post-treatment blood samples will be collected and analyzed for changes in tryptase
Pharmacokinetic Evaluation | From Day 1 to Day 85
  CDX-0159 concentrations will be measured.
Immunogenicity Evaluation | From Day 1 to Day 85
  Patients will be monitored for the development of anti-drug antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany